CLINICAL TRIAL: NCT01863524
Title: Screening for Abdominal Aortic Aneurysm Using a Portable Transthoracic Echocardiography (TTE) Among Patients With Acute Coronary Syndrome in Intensive Cardiac Care Unit.
Brief Title: Screening for Abdominal Aortic Aneurysm Using a Portable Transthoracic Echocardiography Among Patients With Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Mohamed Jabaren, MD, HaEmek Medical Center, Israel
Other Study IDs: emc130152ctil
Record Dates: First submitted 2013-05-14; First posted 2013-05-29 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Acute Coronary Syndrome
Keywords: Abdominal Aortic Aneurysm (AAA),; Echocardiography (TTE),; Acute Coronary Syndrome (ACS); Patients over 65 years old
MeSH Terms: conditions — Acute Coronary Syndrome; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The prevalence of Abdominal Aortic Aneurysm among 65 years old individuals worldwide is 1-2%. when diagnosis is confirmed by abdominal Ultrasound the prevalence is 5.5% in men and 1% in women.

As abdominal aortic aneurysm and coronary heart disease share common risk factors, patients with acute coronary syndrome represent a high risk population in which screening for another atherosclerotic site is recommended.

Patients admitted for ACS undergo routinely TTE. during the same study, TTE may offer the opportunity to evaluate the cardiac morphology and function and to screen for Abdominal Aortic aneurysm. It was reported by different studies that the Sensitivity of this technique was between 91-96% for AAA screening.

In addition, this method is cheap, available and requires only 2-3 minutes to be added to the standard TTE.

we plan to examine patients admitted with ACS in our Intensive Care Unit for screening AAA by TTE in subcostal views in addition to the standard TTE examination.

ELIGIBILITY:
Inclusion Criteria:

* patients over 65 years old with ACS. patients capable of reading, understanding and signing informed concent

Exclusion Criteria:

* suboptimal TTE windows

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 65 years old with ACS admitted in Intensive Cardiac Care Unit, who will be examined by TTE.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2013-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Abdominal aortic diameter measurement of 30 mm or more by portable transthoracic echocardiography, will be defined as abdominal aortic aneurysm. | Average time period of 72 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Jabaren, MD, Principal Investigator — Haemek Medical Center, Afula, Israel
Locations (2):
- Israel (2):
  - HaEmek MC Cardiology depratment, Afula
  - Haemek Medical Center, Afula

IPD SHARING:
Plan to Share IPD: No